CLINICAL TRIAL: NCT04733638
Title: Automated Detection and Volumetric Assessment of Intracerebral Hemorrhage Using Artificial Intelligence- Multicenter Study
Brief Title: ADVANCE- Automated Detection and Volumetric Assessment of ICH
Status: Completed | Type: Observational
Sponsor: Viz.ai, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: Viz-ICH-02
Record Dates: First submitted 2021-01-27; First posted 2021-02-02 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Intracerebral Hemorrhage
Keywords: Artificial Intelligence; ICH
MeSH Terms: conditions — Cerebral Hemorrhage

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Pre-Viz ICH VOLUME: Patient data collected prior to Viz ICH VOLUME implementation, utilized as a control data set
- Post-Viz ICH VOLUME: Patient data collected post-Viz ICH VOLUME implementation
  Interventions: Device: Viz ICH VOLUME

INTERVENTIONS:
Device: Viz ICH VOLUME — Viz ICH VOLUME software is a module that identifies and segments Intraparenchymal Hemorrhage (IPH) from NCCT imaging. This software is for investigational use in the study and is not FDA cleared. For subjects who undergo a brain scan, Viz will use deep learning algorithms to analyze computed tomography (CT) or magnetic resonance (MR) images of the brain for ICH in parallel to standard of care image interpretation. If a suspected ICH is detected, Viz will perform an automatic volumetric analysis and will send a notification to a specialist, such as a neurointerventionalist or a neurosurgeon. Notifications prompt the specialist to review the patient's case. Additionally, non-diagnostic previewing of DICOM images, and HIPAA-compliant text messaging and phone calls are available in the software platform. Viz ICH VOLUME is not intended for use in the diagnosis of disease or other conditions, or in the cure, mitigation, treatment, or prevention of disease, in man.
  Groups: Post-Viz ICH VOLUME

SUMMARY:
To evaluate the performance of the Viz ICH VOLUME algorithm.

DETAILED DESCRIPTION:
To evaluate the performance of the Viz ICH VOLUME algorithm to:

1. detect the presence of ICH on brain imaging,
2. measure the volume of ICH on brain imaging,
3. and to assess the algorithm processing time,
4. and the difference in time to notification, time to treatment, and clinical outcomes in comparison to standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (18 and older)
* Presenting with symptoms suspicious for an acute stroke / intracranial hemorrhage
* Having a complete imaging data set including NCCT +/- MRI, CTA and/or MRA

Exclusion Criteria:

* Subjects with poor or incomplete brain imaging.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive patients, that meet eligibility criteria, undergoing imaging for a suspected acute stroke or intracranial hemorrhage
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2021-01-26 (Actual); Primary Completion 2023-04-15 (Actual); Study Completion 2023-04-28 (Actual)

PRIMARY OUTCOMES:
Algorithm Performance | Up to 10 minutes
  Sensitivity and specificity of Viz ICH VOLUME in detecting ICH compared to standard of care evaluation.

SECONDARY OUTCOMES:
Algorithm Processing Time | Up to 10 minutes
  Total run time in minutes for the algorithm to process the CT scan following receipt
Time to Notification | Up to 10 minutes
  Time in minutes from CT imaging to time an interventionalist was notified
Time to Treatment | up to 1 day (1440 minutes)
  Time in minutes from CT imaging to start time of treatment
Length of Stay | Hospital admit to discharge, up to 30 days
  Number of days in hospital
In Hospital Complications | Hospital admit to discharge, up to 30 days
  Occurrence of stroke-related or stroke treatment-related complications while in hospital
Modified Rankin Scale (mRS) at Discharge and 90 Days | 90 days
  The Modified Rankin Score (mRS) is a 6 point disability scale with possible scores ranging from 0 to 5. A separate category of 6 is usually added for patients who expire. A score of 0 is a patient with no residual symptoms. Scores increase with severity to 5 which equals severe disability.

CONTACTS AND LOCATIONS:
Overall Officials: Moleen Madziva, Study Director — Director of Clinical Affairs at Viz
Locations (5):
- United States (5):
  - Swedish Medical Center Healthone, Englewood, Colorado
  - Mount Sinai Hospital (Neurosurgery), New York, New York
  - Presbyterian Medical Center, Charlotte, North Carolina
  - Forsyth Medical Center, Winston-Salem, North Carolina
  - Prisma Health Upstate, Greenville, South Carolina

IPD SHARING:
Plan to Share IPD: Undecided